CLINICAL TRIAL: NCT04445064
Title: Activity and Safety of Peptide-based Immunotherapy in an Umbrella Window-of-opportunity Phase II Study in Patients With Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Activity and Safety of Peptide-based Immunotherapy in Patients With Squamous Cell Carcinoma of the Head and Neck.
Acronym: HN1901
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unmet primary endpoint
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN1901
Record Dates: First submitted 2020-06-03; First posted 2020-06-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Oropharynx Squamous Cell Carcinoma; Larynx Squamous Cell Carcinoma; Hypopharynx Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma
Keywords: vaccine; immunotherapy; squamous cell carcinoma; head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Intervention Model Description: Multicentric
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: IO102 vaccine (Experimental): Randomization between arm A and B. Patients in arm A will receive IO102 3 to 4 times prior to curative treatment
  Interventions: Biological: IO102
- Arm B: Control group (No Intervention): Randomization between arm A and B
- Arm C: IO103 (Experimental): No randomization. Patients in arm C will receive IO103 3 to 4 times prior to curative treatment
  Interventions: Biological: IO103

INTERVENTIONS:
Biological: IO102 — 100µg each week during the 3 weeks prior to curative treatment (total of 3 to 4 doses maximum)
  Arms: Arm A: IO102 vaccine
Biological: IO103 — 100µg each week during the 3 weeks prior to curative treatment (total of 3 to 4 doses maximum)
  Arms: Arm C: IO103

SUMMARY:
The purpose of this project is to realize a randomized open-label study (EudraCT number: 2020-000120-19) to evaluate the safety and the anti-tumor activity of peptide(s)-based immunotherapy in an umbrella window pre-operative opportunity phase II study in patients with squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Patients with a head and neck squamous cell carcinoma eligible for curative treatment are eligible for this proof of concept study. The included patients in arm A will receive IO102 subcutaneous at 100μg every week during the three weeks following the first endoscopy. The included patients in am B (control group) won't receive any treatment. The included patients in arm C will receive IO103 subcutaneous at 100μg every week during the three weeks following the first endoscopy.

The main objectives of this study are:

* To evaluate the T-cell peptide-specific response to the vaccine in a interferon(INF)-γ ELISpot assay.
* To assess the safety and tolerability of the vaccine.
* To investigate the decreased action of the IDO enzyme in evaluating the increased tumoral infiltration by CD8+ T-lymphocytes and by measuring the serum levels of kynurenin, tryptophan,...
* To evaluate the anti-tumor effect (objective response rate, overall survival, disease free- survival, disease specific survival).
* To evaluate the pre-operative activity of peptide vaccine using MRI (Magnetic Resonance Imaging), DWI-MRI (Diffusion Weighted Imaging-MRI) and MRS (Magnetic Resonance Spectroscopy) to visualize possible significant tumor modifications.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age on day of signing informed consent.
2. Histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx.
3. Patients selected for a surgical treatment.
4. No distant metastases.
5. Measurable disease as per RECIST 1.1.
6. No active second malignancy during the last 3 years except non melanomatous skin cancer or carcinoma in situ of the cervix.
7. The participant provides written signed informed consent for the trial in accordance with ICH-GCP and local legislation prior to admission to the trial.
8. Eastern Cooperative Oncology Group (ECOG) performance status scale 0-1 and Karnofsky score > or = 70.
9. Neutrophil count > 1,500/mm3, platelet count > 75,000/mm3, WBC> or = 3.0/109 L, bilirubin or creatinine < 2 times ULN, ALT or AST < 5 times ULN, Hemoglobin ≥ 9 g/dL.
10. A male participant able to father a child must agree to use contraception starting with the screening visit and throughout the duration of the trial.
11. A female participant is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP).
    2. A WOCBP who agrees to follow contraceptive guidance starting with the screening and throughout the duration of the trial. WOCBP are allowed in the trial if they are using proper contraception (follow guidelines from the European Union Heads of Medicines Agency (CTFG, 2014).

Exclusion Criteria:

1. Nasopharynx cancer, unknown primary and nasal cavity and paranasal sinuses carcinomas.
2. Previous exposure to immunotherapy.
3. Known diagnosis of immune deficiency or a positive serology of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
4. Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) or pre-existing liver cirrhosis.
5. Other uncontrolled active illnesses or nonmalignant systemic disease (examples include, but are not limited to, active infections requiring antibiotics, bleeding disorders, uncontrolled diabetes, uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome).
6. Has received a live vaccine within 30 days prior to the first dose of trial treatment
7. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial treatment.
9. Any psychiatric, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
10. Any malignancy (other than squamous cell carcinoma of the head and neck, non-melanoma skin cancer or localized cervical cancer or localized and presumed cured prostatic cancer or basal cell carcinoma of the skin and carcinoma in situ of the cervix or bladder) within the last 3 years prior to registration.
11. Women of Child Bearing Potential (WOCBP) who has a positive urine pregnancy test (e.g., within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Pregnant woman and women who are expecting to conceive.
13. Breastfeeding women.
14. Patients expected to father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with a T-cell peptide-specific response to the vaccine as assessed by an interferon(INF)-γ ELISpot assay. | 2 years
  ELISpot responses will be considered positive when the numbers of IFN-γ secreting cells will be at least twofold greater than the mean value of the baseline and with a minimum of 50 spots (per 5 × 10^5 peripheral blood mononuclear cell (PBMC) ) detected.

SECONDARY OUTCOMES:
Number of participants experiencing toxicity | 2 years
  Maximum grade of each toxicity and percentage of patients experiencing toxicity as assessed by CTC-NCIv5.0.
  Patients will have blood tests before the second and third administration of the vaccine and 4 weeks after surgery and clinical examinations before each administration of the vaccine and during the 3 months after surgery.
Increase in CD8+ T-cell density (cells/mm2) between tumour biopsies taken before and after treatment, as demonstrated by immunohistochemistry. | 2 years
Objective response rate (ORR) by RECIST Version 1.1 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, Principal Investigator — Insitut de Recherche Expérimentale et Clinique, pôle MIRO
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium